CLINICAL TRIAL: NCT04487691
Title: Autologous Nebulized Platelet Lysate for Post COVID-19 Syndrome
Brief Title: Nebulized PL for Post-COVID-19 Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGX2020-RCT01
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Lysate (Experimental): Inhaled nebulized platelet lysate (PL), 2-ml 1x per day for 8 weeks.
  Interventions: Biological: Nebulized Platelet Lysate
- Saline (Active Comparator): Inhaled nebulized normal sterile saline, 2-ml 1x per day for 8-weeks.
  Interventions: Other: Nebulized Sterile Saline

INTERVENTIONS:
Biological: Nebulized Platelet Lysate — Approximately 520 cc of autologous venous blood (within AABB guideline limits) will be drawn and platelet lysate (PL), maximizing the patients baseline platelet levels (~2-4x baseline) will be produced in a clean room setting using the Regenexx, LLC proprietary lab protocols (PL-M) utilizing a double lysis technique. From that sample, a high growth factor lysate will be created using a double lysis technique, and a sample will be retained to quantify the protein profile of the PL via ELISA quantitative analysis. The PL will be aliquoted into 56 (n=28x2) 2-ml ampules using sterile technique which will then be frozen at -20°C. The patient will unfreeze each ampule and place it into a handheld ultrasonic nebulizer and inhale the platelet lysate following the nebulizer manufacture's protocol until the treatment is completed. The treatment will be applied once a day for 8-weeks.
  Arms: Platelet Lysate
Other: Nebulized Sterile Saline — Approximately 520 cc of autologous venous blood (within AABB guideline limits) will be drawn and donated for research purposes to keep patient blinded to group allocation. Sterile normal saline to mimic the appearance of the platelet lysate will be aliquoted into 56 (n=28x2) 2-ml ampules using sterile technique which will then be frozen at -20°C. The patient will unfreeze each ampule and place it into a handheld ultrasonic nebulizer and inhale the sterile saline following the nebulizer manufacture's protocol until the treatment is completed. The treatment will be applied once a day for 8-weeks.
  Arms: Saline

SUMMARY:
To evaluate and compare nebulized platelet lysate to placebo control of saline administered via handheld nebulizer 1x daily for eight weeks to determine effect on lung function in patients with post-COVID-19 ARDS syndrome.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo controlled single-center study using nebulized platelet lysate compared to placebo control of saline administered via handheld nebulizer 1x daily for eight weeks to determine effect on lung function in patients with post-COVID-19 ARDS syndrome.

20 patients randomized to Treatment group: Inhaled nebulized platelet lysate (PL) 1x daily for eight weeks 20 patients randomized to Control group: Inhaled nebulized saline, 1x daily for eight weeks.

Outcomes will be measured at 4-weeks, 8-weeks, 3-months, 6- months

Goals for this study are as follows:

1. Investigate and compare the efficacy of autologous PL inhaled via handheld ultrasonic nebulizer, 2-ml once per day for 4-weeks compared to saline control (Phase 1), early treatment timepoint.
2. Investigate and compare the efficacy of autologous PL inhaled via handheld ultrasonic nebulizer, 2-ml once per day for 8-weeks compared to saline control (Phase 1), final treatment timepoint.
3. Investigate, compare, and monitor long term function and quality of life through 6-months for treatment arm compared to control.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. At least 4-weeks post ventilator or oxygen dependent ARDS treated for at least 48 hours in the ICU
3. Patient is stable enough to have been discharged home
4. Male or female ages 18-85
5. Two weeks to 1-year post hospital discharge
6. Ongoing activity intolerance due to dyspnea related to ARDS
7. Is independent, ambulatory, and can comply with all post-operative evaluations and visits
8. 6-minute walk test distance of < 450 M
9. SF-36 physical component score < 60
10. ARDS caused by viral pneumonia including COVID-19 confirmed through an RNA anti-body test
11. Normal to mild post-ARDS reactive airway disease

Exclusion Criteria:

1. Oxygen dependent on nasal canula greater than 2-L per minute
2. Dependent on inhaled corticosteroid at the discretion of the physician
3. Unable to complete any of the outcomes measured (Spirometry, 6MWD, SF-36, etc.)
4. Active known secondary bacterial or viral infection
5. Active moderate or severe post-ARDS reactive airway disease at the discretion of the physician
6. Pre-morbid COPD
7. Medication list will be reviewed on a case by case basis to allow for flexibility as post-COVID-19 patients' medication list may vary
8. Other medical comorbidities/conditions that may preclude participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Spirometry-FVC and FEV1/FVC tests | 4 weeks; 8 weeks
  Changes in pre and post treatment spirometry measures

SECONDARY OUTCOMES:
Spirometry-FVC and FEV1/FVC tests | 3 months, 6 months
  Changes from pre and post treatment spirometry measures
6 Minute Walk Distance test (6MWD) | 4 weeks; 8 weeks; 3 months; 6 months
  Changes in distance walked during 6MWD test from pre to post treatment
Distance-desaturation product from 6MWD | 4 weeks; 8 weeks; 3 months; 6 months
  Changes in distance-desaturation product from 6MWD from pre to post treatment
San Diego Shortness of Breath Questionnaire (SOBQ) | 4 weeks; 8 weeks; 3 months; 6 months
  Changes in San Diego Shortness of Breath Questionnaire (SOBQ) score from pre to post; treatment; scores range from 0-120 with higher scores equaling greater breathing impairment
Short Form-36 (SF-36) | 4 weeks; 8 weeks; 3 months; 6 months
  Changes in SF-36 scores from pre to post treatment; 8 subscales 0-100 range where lower scores equal more disability
Modified Single Assessment Numeric Evaluation (SANE) | 4 weeks; 8 weeks; 3 months; 6 months
  Average SANE score post treatment; scores range from 0-100 where 0=no improvement and 100=100% improvement in breathing condition
Medications | 4 weeks; 8 weeks; 3 months; 6 months
  changes in medications from pre to post treatment
Incidence of adverse events | 4 weeks; 8 weeks; 3 months; 6 months
  Incidence of adverse events after treatment
Incidence of surgical/other treatment interventions | 4 weeks; 8 weeks; 3 months; 6 months
  Incidence of surgical/other treatment interventions after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prem K, Liu Y, Russell TW, Kucharski AJ, Eggo RM, Davies N; Centre for the Mathematical Modelling of Infectious Diseases COVID-19 Working Group; Jit M, Klepac P. The effect of control strategies to reduce social mixing on outcomes of the COVID-19 epidemic in Wuhan, China: a modelling study. Lancet Public Health. 2020 May;5(5):e261-e270. doi: 10.1016/S2468-2667(20)30073-6. Epub 2020 Mar 25. PMID 32220655
- [Background] Chan KS, Pfoh ER, Denehy L, Elliott D, Holland AE, Dinglas VD, Needham DM. Construct validity and minimal important difference of 6-minute walk distance in survivors of acute respiratory failure. Chest. 2015 May;147(5):1316-1326. doi: 10.1378/chest.14-1808. PMID 25742048
- [Background] Hopkins RO, Weaver LK, Collingridge D, Parkinson RB, Chan KJ, Orme JF Jr. Two-year cognitive, emotional, and quality-of-life outcomes in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2005 Feb 15;171(4):340-7. doi: 10.1164/rccm.200406-763OC. Epub 2004 Nov 12. PMID 15542793
- [Background] Salama SM, Kamel IH, Ghanim M, Elsherif A. (2019). The Efficacy of Autologous Nebulized Platelet Rich Plasma (PRP) As an Early Adjuvant Therapeutic and Prognostic Treatment Modality in the Management of Inhalation Lung Injury. Egypt, J Plast Reconstr Surg. 43: 203-208. 10.21608/ejprs.2019.65115
- [Background] Geiger S, Hirsch D, Hermann FG. Cell therapy for lung disease. Eur Respir Rev. 2017 Jun 28;26(144):170044. doi: 10.1183/16000617.0044-2017. Print 2017 Jun 30. PMID 28659506
- [Background] Rubio MM. (2019). Beyond the Ordinary: The Effect of Cellular Therapy on Quality of Life in Chronic Lung Disease. J Clin Res Med. 2(4): 1-8. https://researchopenworld.com/beyond-the-ordinary-the-effect-of-cellular-therapy-on-quality-of-life-in-chronic-lung-disease/ Accessed 3/27/20.
- [Background] Mammoto T, Chen Z, Jiang A, Jiang E, Ingber DE, Mammoto A. Acceleration of Lung Regeneration by Platelet-Rich Plasma Extract through the Low-Density Lipoprotein Receptor-Related Protein 5-Tie2 Pathway. Am J Respir Cell Mol Biol. 2016 Jan;54(1):103-13. doi: 10.1165/rcmb.2015-0045OC. PMID 26091161
- [Background] Centeno C, Markle J, Dodson E, Stemper I, Hyzy M, Williams C, Freeman M. The use of lumbar epidural injection of platelet lysate for treatment of radicular pain. J Exp Orthop. 2017 Nov 25;4(1):38. doi: 10.1186/s40634-017-0113-5. PMID 29177632
- [Background] Del Fante C, Perotti C, Bonferoni MC, Rossi S, Sandri G, Ferrari F, Scudeller L, Caramella CM. Platelet lysate mucohadesive formulation to treat oral mucositis in graft versus host disease patients: a new therapeutic approach. AAPS PharmSciTech. 2011 Sep;12(3):893-9. doi: 10.1208/s12249-011-9649-3. Epub 2011 Jul 6. PMID 21732159